CLINICAL TRIAL: NCT06498076
Title: Management of Postspinal Anesthesia Hypotension During Elective Cesarean Section: Baby Norepinephrine Versus Ephedrine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Charles Nicolle (Other)
Responsible Party: Principal Investigator, jebri alia, Head of anesthesia and intensive care departement, Hopital Charles Nicolle
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCharlesNicolle
Record Dates: First submitted 2024-06-13; First posted 2024-07-12 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia Complication; Vasopressor; Cesarean Section Complications; Hypotension During Surgery
Keywords: spinal anesthesia; cesarean section; complications; hypotension; ephedrine; norepinehrine
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine; Ephedrine

STUDY DESIGN:
Intervention Model Description: Groupe N : parturients will received norepinephrine boluses (8 µg) ; prophylactic bolus immediately after spinal anesthesia induction and therapeutic boluses when systolic blood pressure falls to ≤ 20% of baseline.
  Groupe E : parturients will received ephedrine boluses (6 mg) ; systematic bolus after the induction of spinal anesthesia and therapeutic boluses if hypotention.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A total of 126 parturienst are randomly divided into two equal groups by an investigator not directly linked to the study.
  Groupe N : patients will received norepinephrine boluses (8 µg) ; prophylactic bolus immediately after spinal anesthesia induction and therapeutic boluses when systolic blood pressure falls to ≤ 20% of baseline. Groupe E : parturients will received ephedrine boluses (6 mg) ; systematic bolus after the induction of spinal anesthesia and therapeutic boluses if hypotention.
  The syringes will be labeled as syringe A and syringe B and the anesthesiologist who will give the bolus cannot know if it is ephedrine or norepinephrine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group E: ephedrine (Active Comparator): Group E : parturients will received ephedrine boluses (6 mg) ; systematic bolus after the induction of spinal anesthesia and therapeutic boluses if hypotention (systolic blood pressure falls to ≤ 20% of baseline).
  Interventions: Drug: Ephedrine
- Group N: norepinephrine (Active Comparator): Group N : patients will received norepinephrine boluses (8 µg) ; prophylactic bolus immediately after spinal anesthesia induction and therapeutic boluses when systolic blood pressure falls to ≤ 20% of baseline
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — injection of prophylactic norepinephrinebolus after spinal anesthesia induction. If hypotension at any time during surgery, administration of rescue bolus of the same vasopressor to each patient.
  Other Names: Group N
  Arms: Group N: norepinephrine
Drug: Ephedrine — injection of prophylactic ephedrine If hypotension at any time during surgery, administration of rescue bolus of the same vasopressor to each patient.
  Other Names: Group E
  Arms: Group E: ephedrine

SUMMARY:
Background : Spinal anesthesia emerges as the preferred anesthesia technique for elective cesarean section . It offers a preferable alternative to general anesthesia because it provides better maternal safety and neonatal outcomes. However, spinal anesthesia is not free of inherent risks. Hypotension remains the most common complication which threats both mother and child. The common method of treating hypotension includes fluid loading and the use of vasopressors such as ephedrine and phenylephrine. One promising approach is the administration of diluted norepinephrine. It presents a good alternative to preserve maternal blood pressure while minimizing adverse effects on the mother and fetus. Thus, our study proposes to evaluate the efficacy and safety of diluted norepinephrine boluses compared with ephedrine on the management of post- spinal anesthesia hypotension during scheduled cesarean sections.

Patients and methods : After local Ethical Commitee approval, this prospective randomized double -blind study will be undertaken from August to October 2024 in the Department of Anesthesiology and Intensive care and Gynecology and Obstetric department of Charles Nicolle Hospital of Tunis. After obtaining informed written consent, singleton full-term pregnant females of ASA grade II, aged 18-38 years, scheduled for elective cesarean section under spinal anesthesia will be randomly divided into two groups. Group N : patients receive norepinephrine boluses (8 µg) ; prophylactic bolus immediately after spinal anesthesia induction and therapeutic boluses when systolic blood pressure falls to ≤ 20% of baseline. Group E : parturients receive ephedrine boluses (6 mg) ; systematic bolus after the induction of spinal anesthesia and therapeutic boluses if hypotension. Heart rate, systolic, diastolic and mean blood pressure are monitored. Number of episodes of hypotension and number of vasopressor boluses used in each group are recorded and considered as the primary outcomes of the study. Complication during the surgery as incidence of hypertension, tachycardia, bradycardia, nausea and vomiting are recorded. We also record neonatal APGAR score at 1 minute and five minutes. These parameters are considered as the secondary outcomes of the study.

Statistical study:

Data entry and analysis will be performed by SPSS software version 25.0. We will use Excel 2019 software to edit the charts. Continuous quantitative variables following a normal distribution will be expressed by their means and standard deviation. Categorical variables will be expressed as frequencies and percentages. Analytical study: We'll use the Pearson chi2 test or Fischer's exact test, whichever appropriate, for the comparison of categorical variables. T test of Student and Mann Whitney U-test will be employed for comparing Continuous variables. We 'll retain a significance threshold for p less than 5%.

DETAILED DESCRIPTION:
Background : Spinal anesthesia emerges as the preferred anesthesia technique for elective cesarean section . It offers a preferable alternative to general anesthesia because it provides better maternal safety and neonatal outcomes. However, spinal anesthesia is not free of inherent risks. Among the feared complications, hypotension remains the most common complication which threats both mother and child. In this perspective, several preventive and curative means have been studied to optimize maternal and fetal homeostasis. The common methods include fluid loading and the use of vasopressors such as ephedrine and phenylephrine. One promising approach is the administration of diluted norepinephrine. Due to its low agonist activity of the ß receptor and its powerful α adrenergic agonist activity, it presents a good alternative to preserve maternal blood pressure while minimizing adverse effects on the mother and fetus. Thus, our study proposes to evaluate the efficacy and safety of diluted norepinephrine boluses compared with ephedrine on the management of post- spinal anesthesia hypotension during scheduled cesarean sections.

Patients and methods : After approval from the Local Ethical Commitee of the Hospital (N° FWA 00032748) , and after obtaining informed written consent this prospective randomized double -blind study will be undertaken from August to October 2024 in the Department of Anesthesiology and Intensive care and Gynecology and Obstetric department of Charles Nicolle Hospital of Tunis.

Inclusion criteria : Singleton full-term consenting pregnant females of ASA grade II, aged 18-38 years, scheduled for elective cesarean section under spinal anesthesia are included in the study.

Non inclusion criteria : Any parturient falling in the category ASA grade III and IV, contraindications to spinal anesthesia, preeclampsia, chronic hypertension, comorbidity with diabetes mellitus, cardiovascular disorders and psychiatric illness are non included.

Exclusion criteria : They are excluded the case of failure of spinal anesthesia, conversion to general anesthesia, post-partum bleeding, and failure to follow protocol.

Patient groups :

Sample size : It was calculated by (https://statulator.com/SampleSize/ss2M.html), by adjusting a power of 80%, confidence level of 95%, and margin of error of 5%. The primary outcome variable of our study is to compare the number of vasopressor boluses to maintain mean blood pressure ≥ 80% between the groupes, which was estimated from the study conducted by Elnabtity and Selim. The least number of patients required in each groupe with a standard deviation of 2 is 63.

A total of 126 parturients are randomly divided into two equal groups by an investigator not directly linked to the study.

Group N : patients will received norepinephrine boluses (8 µg) ; prophylactic bolus immediately after spinal anesthesia induction and therapeutic boluses when systolic blood pressure falls to ≤ 20% of baseline. Group E : parturients will received ephedrine boluses (6 mg) ; systematic bolus after the induction of spinal anesthesia and therapeutic boluses if hypotension.

The syringes will be labeled as syringe A and syringe B and the anesthesiologist who will give the bolus cannot know if it is ephedrine or norepinephrine.

The preparation of diluted norepinephrine is done by two dilutions: first dilution: 1ml of norepinephrine 2 mg/ml is diluted to 50 ml with 0.9% normal saline to have a concentration of 40 µg/ml. The second dilution: 1ml of norepinephrine 40µg/ml is diluted to 10 ml with 0.9% normal saline in 10 ml syringe prepared as final concentration of 4 µg/ml.

Ephedrine is prepared in 10 ml syringe at a concentration of 3 mg/ml. Preoperative period : A preanesthesia consultation is performed for patients included in the protocol. The modalities of the young preoperative, the anesthetic technique, the protocol of the study are explained to the parturients. Written and signed informed consent by the patients included in the study is obtained.

Intraoperative setting : On arrival to the operating room after a Check list, The parturient is positioned on the operating table in the supine position with left uterine displacement. We use a standard monitoring including non invasive blood pressure (NIBP), pulse oxymeter (SpO2) and electrocardiogram (ECG). We record three values of systolic, diastolic, and mean blood pressure and heart rate before any patient stimulation. An intravenous canula 18 G is inserted and antibiotic prophylaxis is administered 30 minutes before surgical incision using 2 g of cefazolin or 900 mg of clindamycin in case of allergy to penicillins.

Induction of spinal anesthesia: Co fluid loading 10 ml /kg of crystalloids is commenced. In the sitting position, under all aseptic precautions, introduction of spinal needle 25 gauge at L3-L4 or L4-L5 vertebral interspace. After obtaining free flow of cerebrospinal fluid, a standard mixture of anesthetic product : 10 mg of hyperbaric bupivacaine 0.5% (08 mg if parturient's size ≤ 160 cm) with 2.5 µg of sufentanil and morphine 0.1 mg is injected. After intrathecal injection, parturients take quickly their initial position and the first prophylactic bolus of the vasopressor (2 ml) from syringe A or syringe B is administerated. Oxygen is administred by ventimask at rate of 3 l/min till the delivery of the baby. The level of sensory block is evaluated by pin prick test. Successful sensory block is defined as block reaching T4 dermatomal level. If after 20 minutes the sensory block level remains < T10, a conversion to general anesthesia is performed and the patient is excluded from the study.

Heart rate, systolic, diastolic and mean blood pressure are recorded every minute for the first 15 minutes after spinal anesthesia and every five minutes until the end of the intervention.

Management of hypotension : When systolic blood pressure (SBP) decreases to ≤ 20% of baseline, a rescue bolus of vasopressor (2 ml of syringe A or syringe B) is given. Reinjection of the same bolus is repeated after 1 minute if hypotension persists. Administration of boluses is stopped when the value of the SBP finds ≥ 80% of the baseline.

After clamping of the umbilical cord, Oxytocin is given as an initial bolus of 10 UI over 3 minutes followed by slow infusion of 15 UI in 0.9% normal saline. Neonatal APGAR score at 1 minute and five minutes is recorded.

Primary outcome : Number of vasopressor boluses used in each group to treat hypotension (SBP decreases to ≤ 20% of baseline) is recorded.

Secondary outcomes : Complication during the surgery as incidence of hypertension (SBP ≥ 20% of baseline), tachycardia (Heart rate ; HR ≥ 120 beats/min), bradycardia (HR ≤ 60 beats/min), nausea and vomiting are recorded. We'll also recorded neonatal APGAR score of the first and 5th minute.

Statistical study:

Data entry and analysis will be performed by SPSS version 25.0 software We will use Excel 2019 software to edit the charts. Descriptive study: Continuous quantitative variables following a normal distribution will be expressed by their means and standard deviation. Continuous quantitative variables not following a normal law will be expressed by their median and interquartile [25%-75%]. Qualitative variables will be expressed as simple frequencies (n) and relative frequencies as a percentage. Analytical study: For the analysis of the association between two qualitative variables, we will use the Pearson chi-2 test for the comparison of two frequencies under verified application conditions and the Fischer test otherwise. For the analysis of the association between a qualitative variable and a quantitative variable, we 'll use the T test of Student for the comparison of two means and the non-parametric test of Mann Whitney otherwise. We 'll retain a significance threshold for p 5%. In the multivariate study, risk will be calculated by the Odds Ratio (OR) with a retained confidence interval of 95% (95% CI).

ELIGIBILITY:
Inclusion Criteria:

* Singleton full-term consenting pregnant females of ASA grade II, aged 18-38 years, scheduled for elective cesarean section under spinal anesthesia

Exclusion Criteria:

* Any parturient falling in the category ASA grade III and IV, contrindications to spinal anesthesia, preeclampsia, chronic hypertension, comorbidity with diabetes mellitus, cardiovascular disorders and psychiatric illness are non included.

They are excluded the case of failure of spinal anesthesia, conversion to general anesthesia, post-partum bleeding, and failure to follow protocol.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
number of boluses of vasopressor during surgery | number of boluses in the first hour after spinal anesthesia
  number of boluses of norepinephrine in Group N and number of boluses of ephedrine in Group E, to maintain systolic blood pressure more than 80% of the baseline

SECONDARY OUTCOMES:
Incidence of hypertension | number of hypertension in the first hour after spinal anesthesia
  Hypertension is defined as systolic blood pressure ≥ 20% of baseline
Incidence of tachycardia | number of tachycardia in the first hour after spinal anesthesia
  tachycardia : Heart Rate ≥ 120 beats/min
Incidence of bradycardia | number of bradycardia in the first hour after spinal anesthesia
  bradycardia : Heart Rate ≤ 60 beats/min)
Incidence of nausea and vomiting | the first hour after spinal anesthesia
  Nausea vomiting is recorded in each group
Neonatal APGAR score | the first hour
  Neonatal APGAR score is recorded at 1 minute and five minutes

CONTACTS AND LOCATIONS:
Overall Officials: Alia Jebri, MD, Study Director — Charles Nicolle Hospital Tunis
Locations (1):
- Charles Nicolle Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mancuso A, De Vivo A, Giacobbe A, Priola V, Maggio Savasta L, Guzzo M, De Vivo D, Mancuso A. General versus spinal anaesthesia for elective caesarean sections: effects on neonatal short-term outcome. A prospective randomised study. J Matern Fetal Neonatal Med. 2010 Oct;23(10):1114-8. doi: 10.3109/14767050903572158. PMID 20088721
- [Background] Sklebar I, Bujas T, Habek D. SPINAL ANAESTHESIA-INDUCED HYPOTENSION IN OBSTETRICS: PREVENTION AND THERAPY. Acta Clin Croat. 2019 Jun;58(Suppl 1):90-95. doi: 10.20471/acc.2019.58.s1.13. PMID 31741565
- [Background] Mercier FJ, Bonnet MP, De la Dorie A, Moufouki M, Banu F, Hanaf A, Edouard D, Roger-Christoph S. [Spinal anaesthesia for caesarean section: fluid loading, vasopressors and hypotension]. Ann Fr Anesth Reanim. 2007 Jul-Aug;26(7-8):688-93. doi: 10.1016/j.annfar.2007.05.003. Epub 2007 Jun 27. French. PMID 17590565
- [Background] Ngan Kee WD, Khaw KS. Vasopressors in obstetrics: what should we be using? Curr Opin Anaesthesiol. 2006 Jun;19(3):238-43. doi: 10.1097/01.aco.0000192816.22989.ba. PMID 16735804
- [Background] Heesen M, Stewart A, Fernando R. Vasopressors for the treatment of maternal hypotension following spinal anaesthesia for elective caesarean section: past, present and future. Anaesthesia. 2015 Mar;70(3):252-7. doi: 10.1111/anae.13007. Epub 2015 Jan 13. No abstract available. PMID 25583307
- [Background] Mohta M, Dubey M, Malhotra RK, Tyagi A. Comparison of the potency of phenylephrine and norepinephrine bolus doses used to treat post-spinal hypotension during elective caesarean section. Int J Obstet Anesth. 2019 May;38:25-31. doi: 10.1016/j.ijoa.2018.12.002. Epub 2018 Dec 13. PMID 30685301
- [Background] Ali Elnabtity AM, Selim MF. Norepinephrine versus Ephedrine to Maintain Arterial Blood Pressure during Spinal Anesthesia for Cesarean Delivery: A Prospective Double-blinded Trial. Anesth Essays Res. 2018 Jan-Mar;12(1):92-97. doi: 10.4103/aer.AER_204_17. PMID 29628561
- [Result] Reynolds F, Seed PT. Anaesthesia for Caesarean section and neonatal acid-base status: a meta-analysis. Anaesthesia. 2005 Jul;60(7):636-53. doi: 10.1111/j.1365-2044.2005.04223.x. PMID 15960713

DOCUMENTS (2):
  • Study Protocol (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT06498076/Prot_000.pdf
  • Informed Consent Form (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT06498076/ICF_001.pdf